CLINICAL TRIAL: NCT05346783
Title: A Phase 1/2. Multicenter, Randomized, Double-blinded, Placebo and Active-controlled, Parallel Study for Comparing Efficacy and Safety of TJO-083 in Dry Eye Disease Patients
Brief Title: Comparing Efficacy and Safety of TJO-083 in Dry Eye Disease Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJO-083-121
Record Dates: First submitted 2022-03-23; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2021-10

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TJO-083 [Part 2] (Experimental): 1 drop 3 times a day
  Interventions: Drug: TJO-083
- Placebo of TJO-083 [Part 2] (Placebo Comparator): 1 drop 6 times a day
  Interventions: Other: Placebo (vehicle)
- Diquas-s Ophthalmic solution 3% 0.4mL [Part 2] (Active Comparator): 1 drop 6 times a day
  Interventions: Drug: Diquafosol ophthalmic sodium solution 3%

INTERVENTIONS:
Drug: TJO-083 — Diquafosol ophthalmic sodium solution, 1 drop 3 times a day
  Arms: TJO-083 [Part 2]
Other: Placebo (vehicle) — 1 drop 6 times a day
  Arms: Placebo of TJO-083 [Part 2]
Drug: Diquafosol ophthalmic sodium solution 3% — Diquafosol ophthalmic sodium solution, 1 drop 6 times a day
  Arms: Diquas-s Ophthalmic solution 3% 0.4mL [Part 2]

SUMMARY:
This is a prospective randomized study compared with active control and placebo arms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 20 or over
* Patient who have been diagnosed with dry eye syndrome at least 6 months ago
* Screening both eyes, the corrected visual acuity is 0.2 or more
* Written informed consent to participate in the trial

Exclusion Criteria:

* Screening visits within 2 months the patients with systemic or ocular disorders affected the test results (ocular surgery, trauma, or disease)
* Intraocular pressure(IOP)> 21 mmHg

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of TJO-083 to use questionnaire [Part1] | Baseline and Day 2, 8
  Changes from Baseline in tolerability questionnaire in 4 point scale at Day 2, 8. The including lists are below.
  Stinging/Burning, Itching, Blurred vision, Sandiness/Grittiness, Dryness, Light sensitivity, Pain or soreness, Hyperemia.
Change From Baseline in Corneal Staining in 9 point Score at Week 4 [Part 2] | Baseline and Week 4
  Change from Baseline in corneal staining of the worse eye using blue fluorescein staining procedure in 9 point scare at Week 4. (As the score high, the condition of eye is worse)

SECONDARY OUTCOMES:
Change From Baseline in Non-anesthetic Schirmer Test at Week 2, 4, 8, 12 [Part 2] | Baseline and Week 2, 4, 8 and 12
  The Schirmer test without anesthesia was used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Keun Lee, MD, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Hyung Keun, Lee, Seoul, South Korea